CLINICAL TRIAL: NCT01282203
Title: Evaluation of VIMA With SEVOrane in Adult Patients Required General Anesthesia fOr Surgery in TErms of Quality of Anesthesia and Its Influence on Cardiovascular sysTem In commON Clinical Practice (SEVOPROTECTION)
Brief Title: Evaluation of Volatile Induction and Maintenance Anesthesia (VIMA) With Sevorane in Adult Patients Required General Anesthesia for Surgery in Terms of Quality of Anesthesia and Its Influence on Cardiovascular System in Common Clinical Practice
Acronym: SEVOPROTECTION
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-638
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-01

CONDITIONS: Anesthesia, General
Keywords: General surgery; General anesthesia; Inhalation anesthesia; Sevorane; Sevoflurane

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adults requiring anesthesia for surgery: This post-marketing observational study will be conducted in a prospective, multi-centre format. It is a non-interventional, observational study in which Sevorane is prescribed for adult patients undergoing general surgery for induction and maintenance of anesthesia in the usual manner in accordance with the terms of the local marketing authorization. Sevorane is used for induction and maintenance anesthesia by the choice of anesthesiologist. No additional procedures (other than standard of care) shall be applied to the patients. Each patient will be observed from the start of anesthesia through anesthesia end. Markers of myocardial ischemia will be detected up to the first 24 hours after anesthesia (if available). Additionally the correlation between the experience and training background of anesthesiologists and patient related outcomes of general anesthesia with Sevorane as a single anesthetic will be assessed.

SUMMARY:
The main objective of this post-marketing observational study is to collect data from the use of general anesthesia in patients undergoing any surgery to create local recommendations. These data will be based on the evaluation of volatile induction and maintenance anesthesia (VIMA) with Sevorane® (sevoflurane) in adult patients requiring general anesthesia for surgery in terms of quality of anesthesia and its influence on cardiovascular system in common clinical practice in Kazakhstan.

DETAILED DESCRIPTION:
This post-marketing observational study will be conducted in a prospective, multi-centre format. It is a non-interventional, observational study in which Sevorane is prescribed for adult patients undergoing general surgery for induction and maintenance of anesthesia in the usual manner in accordance with the terms of the local marketing authorization. Sevorane is used for induction and maintenance anesthesia by the choice of anesthesiologist. No additional procedures (other than standard of care) shall be applied to the patients. Each patient will be observed from the start of anesthesia through anesthesia end. Markers of myocardial ischemia will be detected up to the first 24 hours after anesthesia (if available). Additionally the correlation between the experience and training background of anesthesiologists and patient related outcomes of general anesthesia with Sevorane as a single anesthetic will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing general anesthesia for planned or urgent surgery for whom Sevorane is used for induction and maintenance anesthesia by the choice of anesthesiologist
* Age greater than or equal to 18 years

Exclusion Criteria:

* Known sensitivity to sevoflurane or other anesthetic containing halogen
* Known or suspected genetic susceptibility to malignant hyperthermia
* Receiving regional anesthetic techniques
* Receiving intravenous anesthesia
* A history of unexplained moderate/severe hepatic dysfunction with jaundice, fever, and/or eosinophilia in association with halogenated anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing planned or urgent surgery
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galyna Bryn, PhD, Study Director — Abbott Laboratories S.A., Ukraine
Locations (12):
- Kazakhstan (12):
  - Site Reference ID/Investigator# 51851, Almaty
  - Site Reference ID/Investigator# 54703, Almaty
  - Site Reference ID/Investigator# 51843, Astana
  - Site Reference ID/Investigator# 51844, Astana
  - Site Reference ID/Investigator# 54705, Astana
  - Site Reference ID/Investigator# 51842, Kokshetau
  - Site Reference ID/Investigator# 51847, Kostanay
  - Site Reference ID/Investigator# 64462, Kyzylorda
  - Site Reference ID/Investigator# 54704, Oral
  - Site Reference ID/Investigator# 51845, Semey
  - Site Reference ID/Investigator# 51848, Shymkent
  - Site Reference ID/Investigator# 44446, Zhezqazghan

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults Requiring Anesthesia for Surgery: Adult patients requiring general anesthesia for surgery
Period: Overall Study
Arm/Group | Adults Requiring Anesthesia for Surgery
Started | 1122
Completed | 1121
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1122
Age Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 619
  Male | 503

OUTCOME MEASURES:

1. Primary Outcome: Time to Loss of Consciousness of Patients Administered Anesthesia
Description: Loss of consciousness was measured from the time the anesthetic was administered until loss of consciousness (loss of eyelash reflex) occurred.
Time Frame: Up to 10 minutes
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 945
Minutes | 2.7 (1.4)

2. Primary Outcome: Time to Awakening of Patients
Description: Measured from the time anesthesia administration was stopped until the patient responded to a verbal command.
Time Frame: Every minute after anesthesia was stopped until the patient responded to a verbal command.
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1116
Minutes | 15.4 (19.8)

3. Primary Outcome: Time to Extubation of Patients
Description: Time to extubation was measured from the time anesthesia administration was stopped until tracheal extubation occurred.
Time Frame: Every minute after anesthesia was stopped until extubation occurred
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1010
Minutes | 65.7 (127.5)

4. Primary Outcome: Anesthesiologists' Satisfaction With Using Sevorane for Induction and Maintenance Anesthesia
Description: The overall satisfaction of the anesthesiologist with the inhalation anesthesia with Sevorane for each patient was assessed by means of a numerical rating scale ranging from 0 (dissatisfied) to 10 (very satisfied).
Time Frame: Day 1
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1116
units on a scale | 9.2 (1.1)

5. Primary Outcome: Patients' Overall Impression of Anesthesia With Sevorane
Description: After awakening from anesthesia, patients were surveyed regarding their overall impression of anesthesia with Sevorane. Patients selected one of the following answers: Excellent, positive, indifferent, or other.
Time Frame: Day 1
Population: All participants with available data were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1114
Participants
  Excellent | 476
  Positive | 627
  Indifferent | 11
  Other | 0

6. Secondary Outcome: Systolic Blood Pressure
Description: The systolic blood pressure of each patient was recorded at different time points from just before the start of anesthesia to one hour after the surgery concluded.
Time Frame: Before starting anesthesia to one hour after the surgery
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 995
mm Hg
  Before anesthesia | 137.5 (23.9)
  Induction anesthesia (after intubation) | 125.3 (22.3)
  After surgical incision | 117.6 (17.8)
  After extubation | 125.5 (14.1)
  One hour after surgery | 124.2 (12.5)

7. Secondary Outcome: Diastolic Blood Pressure
Description: The diastolic blood pressure of each patient was recorded at different time points from just before the start of anesthesia to one hour after the surgery concluded.
Time Frame: Before starting anesthesia to one hour after the surgery
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 995
mm Hg
  Before anesthesia | 84.7 (13.4)
  Induction anesthesia (after intubation) | 78.5 (30.2)
  After surgical incision | 73.2 (12.3)
  After extubation | 77.9 (11.7)
  One hour after surgery | 76.9 (10.5)

8. Secondary Outcome: Mean Arterial Pressure
Description: The mean arterial pressure of each patient was recorded at different time points from just before the start of anesthesia to one hour after the surgery concluded.
Time Frame: Before starting anesthesia to one hour after the surgery
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 973
mm Hg
  Before anesthesia | 103.9 (17.9)
  Induction anesthesia (after intubation) | 95.3 (18.0)
  After surgical incision | 89.5 (15.0)
  After extubation | 95.5 (13.0)
  One hour after surgery | 95.0 (12.1)

9. Secondary Outcome: Heart Rate
Description: The heart rate of each patient was recorded at different time points from just before the start of anesthesia to one hour after the surgery concluded.
Time Frame: Before starting anesthesia to one hour after the surgery
Population: All participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 983
beats per minute
  Before anesthesia | 83.4 (14.9)
  Induction anesthesia (after intubation) | 81.9 (15.0)
  After surgical incision | 79.1 (13.5)
  After extubation | 82.8 (10.4)
  One hour after surgery | 79.2 (9.0)

10. Secondary Outcome: Presence of Deviations in Electrocardiogram Assessments During Anesthesia
Description: Electrocardiogram (ECG) assessments performed during induction of the anesthesia and maintenance were analyzed with respect to the presence of the following deviations: Blockades (problems with heart electrical activity), extrasystoles (extra abnormal heart beats), arrhythmia (abnormal heart rate or rhythm), and myocardial ischemia (decreased blood flow to the heart).
Time Frame: During induction and maintenance of anesthesia
Population: All participants with valid data were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1057
Participants
  Blockades (induction) | 9
  Blockades (maintenance) | 12
  Extrasystoles (induction) | 3
  Extrasystoles (maintenance) | 10
  Arrhythmia (induction) | 8
  Arrhythmia (maintenance) | 21
  Myocardial ischemia (induction) | 70
  Myocardial ischemia (maintenance) | 74

11. Secondary Outcome: Cardiac Troponin (if Available)
Description: Troponin T values measured within 24 hours of anesthesia were to be collected when available.
Time Frame: Within 24 hours after anesthesia
Population: No data were available for the cardiac troponin outcome measure.
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 0

12. Secondary Outcome: Creatine Kinase Myocardial Isoenzyme (if Available)
Description: Creatine kinase myocardial isoenzyme values measured within 24 hours of anesthesia were to be collected when available.
Time Frame: Within 24 hours after anesthesia
Population: No data were available for the creatine kinase myocardial isoenzyme outcome measure.
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 0

13. Secondary Outcome: Correlation Between Anesthesiologists' Clinical Experience and Hemodynamic Parameters During Anesthesia
Description: The anesthesiologists' length of clinical experience with Sevorane was collected (see Outcome Measure 15). The influence of this experience on the changes in hemodynamic parameters during anesthesia with Sevorane was evaluated by calculating Spearman's correlation coefficient between the duration of clinical experience with Sevorane and the changes in blood pressure, mean arterial pressure, and heart rate between T0 (before anesthesia) and T1 (at the end of induction), T2 (at the end of surgical incision), T3 (at the end of extubation), T4 ( 1 hour after the surgery), and the minimum and maximum values, respectively.
Time Frame: Before starting anesthesia to one hour after the surgery
Population: All participants with available data at each time point were included in the analysis.
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1121
Spearman's correlation coefficient
  Systolic blood pressure (T1- T0; n=1121) | 0.271
  Systolic blood pressure (T2-T0; n=1121) | 0.207
  Systolic blood pressure (T3 -T0; n=1005) | 0.143
  Systolic blood pressure (T4 -T0; n=1105) | 0.131
  Systolic blood pressure (Minimum -T0; n=1120) | 0.213
  Systolic blood pressure (Maximum -T0; n=1120) | 0.153
  Diastolic blood pressure (T1-T0; n=1119) | 0.289
  Diastolic blood pressure (T2-T0; n=1119) | 0.243
  Diastolic blood pressure (T3-T0; n=1005) | 0.203
  Diastolic blood pressure (T4-T0; n=1105) | 0.196
  Diastolic blood pressure (Minimum-T0; n=1118) | 0.288
  Diastolic blood pressure (Maximum-T0; n=1118) | 0.163
  Mean arterial blood pressure (T1-T0; n=1101) | 0.308
  Mean arterial blood pressure (T2-T0; n=1102) | 0.250
  Mean arterial blood pressure (T3-T0; n=988) | 0.199
  Mean arterial blood pressure (T4-T0; n=1084) | 0.196
  Mean arterial blood pressure (Minimum-T0; n=1099) | 0.288
  Mean arterial blood pressure (Maximum-T0; n=1099) | 0.177
  Heart rate (T1-T0; n=1117) | 0.269
  Heart rate (T2-T0; n=1116) | 0.245
  Heart rate (T3-T0; n=995) | -0.040
  Heart rate (T4-T0; n=1101) | -0.030
  Heart rate (Minimum-T0; n=1115) | 0.223
  Heart rate (Maximum-T0; n=1116) | 0.120

14. Secondary Outcome: Correlation Between Anesthesiologists' Clinical Experience and Time to Extubation and Awakening
Description: Anesthesiologists' length of clinical experience with general anesthesia and modern inhalation agents was collected (see Outcome Measure 15). The influence of this clinical experience on anesthesia parameters was evaluated by calculating Spearman's correlation coefficient between the duration of clinical experience with inhalation anesthesia and Sevorane on the time to extubation and the time to awakening, respectively.
Time Frame: Every minute after anesthesia was stopped until the patient was extubated and until the patient responded to a verbal command
Population: All participants with available data at each time point were included in the analysis.
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Adults Requiring Anesthesia for Surgery
Number analyzed (Participants) | 1116
Spearman's correlation coefficient
  Exp w/ inh anesthesia (time to extubation; n=1010) | -0.720
  Exp w/ inh anesthesia (time to awakening; n=1116) | -0.415
  Exp w/ Sevorane (time to extubation; n=1010) | -0.681
  Exp w/ Sevorane (time to awakening; n=1116) | -0.294

15. Secondary Outcome: Anesthesiologists' Duration of Clinical Experience With Anesthesia
Description: Mean number of years of participating anesthesiologists' clinical experience with general anesthesia, with modern inhalation agents, and with Sevorane. (See Outcome Measures 13 and 14 for correlated data.)
Time Frame: Baseline
Population: Number of anesthesiologists participating in study.
Measure: Mean (Standard Deviation); unit: years
Groups:
- General Anesthesia: Duration of experience with general anesthesia.
- Inhalation Anesthesia: Duration of experience with inhalation anesthesia.
- Anesthesia With Sevorane: Duration of experience with Sevorane.
Arm/Group | General Anesthesia | Inhalation Anesthesia | Anesthesia With Sevorane
Number analyzed (Participants) | 12 | 12 | 12
years | 17.8 (9.2) | 15.4 (11.6) | 3.5 (2.5)

ADVERSE EVENTS:
Time Frame: Physicians reported all serious adverse events occurring during the induction, maintenance, and recovery phases of surgery until 30 days or 5 half-lives following termination of Sevorane. Mean (SD) total duration of anesthesia was 98.4 (67.2) minutes.
Arm/Group | Adults Requiring Anesthesia for Surgery
Serious Adverse Events (participants affected / at risk) | 4/1122
Other Adverse Events (participants affected / at risk) | 1/1122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults Requiring Anesthesia for Surgery (N=1122)
Ventricular fibrillation (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 1
Hypokalemia (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults Requiring Anesthesia for Surgery (N=1122)
Blood pressure increased (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Troponin T and CK-MB values were not collected in the study, therefore no conclusions can be made regarding the influence of volatile induction and maintenance anesthesia with Sevorane on myocardial ischemia markers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.